CLINICAL TRIAL: NCT00831727
Title: Examining Potential Moderators and Mediators in the Expressive Writing Intervention: The Role of Affect Regulation and Self-presentation.
Brief Title: The Role of Affect Regulation and Self-presentation in the Expressive Writing Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Responsible Party: Principal Investigator, Justin Mattina, Principal Investigator, University of Toronto
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 23614; SSHRC 767-2007-2210-4
Record Dates: First submitted 2009-01-28; First posted 2009-01-29 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-05

CONDITIONS: Posttraumatic Stress Disorders
Keywords: expressive writing; trauma; intervention; posttraumatic stress
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Wounds and Injuries

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Expressive Writing (Experimental)
  Interventions: Behavioral: Expressive Writing
- Control (Placebo Comparator)
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Expressive Writing — Participants will write about their experienced trauma for 20 minutes on each of three consecutive days using techniques associated with expressive writing
  Other Names: Emotional writing
  Arms: Expressive Writing
Behavioral: Control — Participants will write as factually as possible about an assigned trivial topic for 20 minutes on each of three consecutive days
  Arms: Control

SUMMARY:
The purpose of the present study is twofold. First, we will attempt to examine the role that emotion regulation and self-presentation play as potential moderators in the expressive writing paradigm. We hypothesize that expressive writing participants who demonstrate greater abilities to regulate their emotions at baseline will improve more on our outcome measures. We also hypothesize that those expressive writing participants who demonstrate higher levels of self-presentation at baseline will improve less on our outcome measures.

The second aim of the study has two related objectives. First, we will attempt to investigate whether the expressive writing intervention can increase and enhance an individual's emotion regulation abilities. Related to this, we will then go on to examine whether emotion regulation can be looked at as a potential mechanism of action in the expressive writing procedure. Related to these two objectives, we hypothesize that in comparison to the control group, participants in the expressive writing condition will show increases in their ability to regulate their emotions from baseline to four week follow up. Moreover, we predict that greater gains in emotion regulation abilities for the expressive writing participants will be significantly related to greater gains in outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* Fluent in English
* Previously experienced trauma (not current or ongoing; excluding bereavement)
* Currently experiencing trauma-related distress

Exclusion Criteria:

* Currently involved in psychotherapy
* Currently taking psychotropic medications
* Imminent threat to self or others

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2009-02; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Posttraumatic Stress Diagnostic Scale | Initial session; One month follow-up

SECONDARY OUTCOMES:
Difficulties in Emotion Regulation Scale | Initial session; One month follow-up
Pennebaker Inventory of Limbic Languidness | Initial session; One month follow-up
Beck Depression Inventory, Second Edition | Initial session; One month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Jeanne C Watson, Ph.D., Study Director — University of Toronto; Justin M Mattina, M.A., Principal Investigator — University of Toronto; Jonathan J Danson, B.A., Principal Investigator — University of Toronto
Locations (1):
- Ontario Institute for Studies in Education of the University of Toronto, Toronto, Ontario, Canada